CLINICAL TRIAL: NCT03871868
Title: Vitamin D Levels İn Women With and Without Myoma Uteri
Brief Title: Vitamin D Levels And Myoma Uteri
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, pınar kadiroğulları M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2018/11/43
Record Dates: First submitted 2019-03-11; First posted 2019-03-12 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Myoma;Uterus; Vitamin D Deficiency; Polycystic Ovary
Keywords: 25-hydroxyvitamin D
MeSH Terms: conditions — Myofibroma; Vitamin D Deficiency; Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: In Woman With Myoma Uteri
- control group: In Woman Without Myoma Uteri

SUMMARY:
Women with at least one uterine leiomyoma and polycystic ovary syndrome over 10 mm and women with normal ultrasonographic findings were included in the study. Blood samples were taken for biochemical analysis such as vitamin D, calcium, magnesium, phosphorus, thyroid stimulating hormone (TSH), hemoglobin (hb), hematocrit (htc), platelet (plt), and albumin. The study groups were compared in terms of these biochemical markers and family history of patients, daily sunshine hours, clothing preferences and education level.

ELIGIBILITY:
Inclusion Criteria: The reproductive age women (25-50 years) with at least one 10 mm or larger diameter leiomyoma detected by transvaginal ultrasound were the study group.

Exclusion Criteria:

* Patients with a history of myomectomy,
* chronic systemic disease
* malignancy
* history of adenomyosis
* women in menopause
* pregnant women
* vitamin D supplementation
* lactation
* abortion and pregnancy loss in the last 6 months
* oral contraceptive / hormonal agents in the last 3 months

Ages: 25 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — 25-50 years old women with and without myoma uteri
Study Population: The reproductive age women (25-50 years) with at least one 10 mm or larger diameter leiomyoma detected by transvaginal ultrasound were the study group.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Vitamin D levels | december 2018- march 2019
  Vitamin D levels in blood test

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)